CLINICAL TRIAL: NCT04349436
Title: An Open-Label, Multicenter, Phase 1B/2 Study of RP1 in Solid Organ and Hematopoietic Cell Transplant Recipients With Advanced Cutaneous Malignancies
Brief Title: A Phase 1B/2 Study of RP1 in Solid Organ Transplant Patients With Advanced Cutaneous Malignancies
Acronym: ARTACUS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPL-003-19
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma; Basal Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Merkel Cell; Carcinoma, Basal Cell; Melanoma | interventions — MAPRE1 protein, human

STUDY DESIGN:
Intervention Model Description: RP1 injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP1, intra-tumoral injection, oncolytic virus (Experimental): RP1 administered as an intra-tumoral injection every 2 weeks.
  Interventions: Biological: RP1, intra-tumoral injection, oncolytic virus

INTERVENTIONS:
Biological: RP1, intra-tumoral injection, oncolytic virus — Genetically modified herpes simplex type 1 virus

SUMMARY:
This Phase 1B/2 study is a multicenter, open-label, study of RP1 to investigate the (a) objective response rate, in addition to (b) safety and tolerability of RP1 for the treatment of advanced cutaneous malignancies in up to 65 evaluable organ transplant recipients. This will include patients with either previous renal, hepatic, heart, lung, or other solid organ transplantation or hematopoietic cell transplant and experiencing subsequent documented locally advanced or metastatic cutaneous malignancies. The study will enroll a total of 65 evaluable patients. Patients will participate up to approximately 3 years including a 28-day screening period, up to approximately 1 year treatment period, and a 2-year follow-up period.

DETAILED DESCRIPTION:
RP1 is a genetically modified herpes simplex type 1 virus that is designed to directly destroy tumors and to generate an anti-tumor immune response. This is a Phase 1B/2, open label, multicenter, trial evaluating the objective response rate and the safety and tolerability, biodistribution, shedding, and preliminary efficacy of RP1 in adult hepatic, renal, heart, lung, other solid organs, or hematopoietic cell transplant recipients who subsequently experienced advanced or metastatic cutaneous malignancies. Patients will be dosed with RP1 by direct or ultrasound guided intra-tumoral injection into superficial, subcutaneous or nodal tumors. No transplanted organs will be injected.

ELIGIBILITY:
Key Inclusion Criteria:

1. Voluntary agreement to provide written informed consent prior to any study procedures and the willingness and ability to comply with all aspects of the protocol and understand the risk to their organ allograft.
2. Patients with histologically or cytologically confirmed recurrent, locally advanced or metastatic (to skin, soft tissue or lymph nodes) cutaneous malignancies, including CSCC, basal cell carcinoma, Merkel cell carcinoma, and melanoma
3. Patients must have progressed following local resection, prior radiation, topical or systemic therapies.
4. Documentation from the patient's transplant physician confirming that the patient's allograft is stable.
5. Patients for whom surgical or radiation treatment of lesions is contraindicated.
6. At least 1 lesion that is measurable and injectable by study criteria (tumor of ≥1cm in longest diameter or ≥1.5 cm in shortest diameter for lymph nodes).
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
8. Anticipated life expectancy > 6 months
9. Baseline ECG without evidence of acute ischemia.
10. All patients must consent to provide archived or newly obtained tumor material (either formalin-fixed, paraffin-embedded [FFPE] block or 20 unstained slides).

Key Exclusion Criteria:

1. Prior treatment with an oncolytic therapy.
2. Patients with visceral metastases.
3. Patients with active herpetic infections or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis).
4. Patients with a history of organ graft rejection within 12 months.
5. Had systemic infection requiring intravenous (IV) antibiotics or anti-virals, or other serious infection within 60 days prior to dosing.
6. Patients who require intermittent or chronic use of systemic (oral or intravenous) anti-virals with known anti-herpetic activity (e.g., acyclovir) unless for organ allograft preservation.
7. Patients requiring CTLA-4-Ig medications.
8. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments beyond that required for maintenance allograft rejection prevention. The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that requires only hormone replacement, or psoriasis that does not require systemic treatment.
9. Active infection with hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
10. Any history of transplant-related viral infections, such as BKV, EBV or CMV, within 3 months of study entry. Patients with a history of hepatitis B or C virus must have undetectable viral load within 3 months of study entry.
11. Patients with a condition requiring an increase in the patient's usual immunosuppressive medications within 60 days of study treatment.
12. Known active CNS metastases and/or carcinomatous meningitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome Measure | 36 months
  Assess the safety and tolerability of single-agent RP1 in solid organ transplant patients with cutaneous malignancies by incidence of subjects with treatment-emergent adverse events
Primary Efficacy Outcome Measure | 36 months
  The objective response rate (ORR) according to investigator assessment using modified RECIST version 1.1.
Incidence of subjects with treatment-emergent adverse events greater than or equal to Grade 3 | 36 months
Incidence of subjects with Serious adverse events (SAEs) | 36 months
Incidence of subjects with fatal adverse events | 36 months
Treatment-emergent adverse events requiring withdrawal from IP and incidence of organ allograft rejection | 36 months

SECONDARY OUTCOMES:
Duration of response (DOR) by investigator among subjects who experience Complete Response (CR) or Progressive Disease (PD) | 36 months
CR rate by investigator assessment | 36 months
Disease control rate (DCR) by investigator review | 36 months
Clinical benefit rate defined as the rate of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) | 36 months
Progression Free Survival (PFS) by investigator review Duration of clinical benefit (DOCB) during active treatment and for up to one year after last treatment by investigator review | 36 months
Overall survival (OS) at one year and two years | 36 months
3-year survival rate of subjects | 36 months
Quality of life (QoL), as determined by patient-reported outcomes | 36 months
Biologic activity as assessed by changes in individual tumor sizes, erythema, inflammation and necrosis | 36 months
  Percentage of patients with biopsy-proven clinical rejection and percentage of patients who require an increase in immune suppressive therapy, during active treatment and for up to 1 year after last treatment
Disease-free Survival | 36 months
To asses the efficacy of RP1 as determined by ORR in all transplant recipients treated, by investigator review | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: May Cho, MD, Study Director — Replimune Inc.
Locations (28):
- United States (28):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - UCSF, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center School of Medicine, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Rochester Dermatologic Surgery, New York, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center at Knoxville, Knoxville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia